CLINICAL TRIAL: NCT07090278
Title: Ulinastatin Treatment Reduces the Incidence of Sepsis-associated Encephalopathy
Status: Completed | Type: Observational
Sponsor: Shusheng Li (Other)
Responsible Party: Sponsor-Investigator, Shusheng Li, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: SAE-UTI
Record Dates: First submitted 2025-07-15; First posted 2025-07-29 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Sepsis-Associated Encephalopathy
Keywords: sepsis; sepsis-associated encephalopathy; ulinastatin
MeSH Terms: conditions — Sepsis-Associated Encephalopathy; Sepsis | interventions — urinastatin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — In the prospective cohort, the remaining blood after blood routine or arterial blood gas analysis was quickly centrifuged to separate plasma. Plasma samples were immediately stored at -80°C in a dedicated biobank for subsequent batch analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ulinastatin Group: Patients diagnosed with sepsis who received ulinastatin as part of routine clinical care. The use of ulinastatin was not assigned by study protocol but determined by treating physicians. Clinical outcomes, including the incidence of SAE, were assessed.
  Interventions: Drug: ulinastatin
- Non-Ulinastatin Group: Patients diagnosed with sepsis who did not receive ulinastatin treatment during hospitalization. Clinical outcomes, including the incidence of SAE, were recorded. No study-specific interventions were applied.

INTERVENTIONS:
Drug: ulinastatin — Ulinastatin for the treatment of sepsis patients during ICU stay
  Groups: Ulinastatin Group

SUMMARY:
This study was conducted to explore the association between ulinastatin treatment and the incidence of sepsis-associated encephalopathy (SAE) in patients with sepsis. The study was divided into two phases: first, a multicenter retrospective observational cohort: to evaluate the correlation between ulinastatin treatment and the risk of SAE; second, a single center prospective observational cohort: to further explore the association between ulinastatin treatment and SAE.

DETAILED DESCRIPTION:
This study consisted of two parts: a retrospective, multicenter observational derivation cohort and a prospective, single-center observational validation cohort. Both parts of the study included adult patients admitted to the intensive care unit of Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology. The first part of the study, being retrospective in nature, was exempted from obtaining informed consent. However, all participants in the second part of the study signed a written informed consent form. The first part of the study retrospectively collected adult patients with sepsis according to the inclusion and exclusion criteria, explored the factors related to sepsis-related encephalopathy, and analyzed the correlation between the use of ulinastatin treatment and the occurrence of SAE. The second part of the study was a prospective study. After signing the informed consent form, eligible patients were included. After collecting blood routine or arterial blood gas analysis, the remaining blood was centrifuged and the plasma was frozen at -80°C for subsequent detection of nitric oxide.

The primary exposure variable was the administration of ulinastatin in patients with sepsis. Demographic data, including age and gender, were collected at ICU admission. Additional exposure variables included blood biochemical markers and infection-related indicators. Clinical comorbidities were recorded based on established diagnoses documented in the medical record, including hypertension, coronary artery disease, atrial fibrillation, diabetes, respiratory diseases (chronic obstructive pulmonary disease, asthma, chronic bronchitis, and bronchiectasis), renal dysfunction, history of tumor, history of stroke, and liver cirrhosis.

The primary outcome was the occurrence of SAE within 3 days of enrollment. Secondary outcomes in the prospective cohort included the fasting blood glucose/ high density lipoprotein cholesterol (FBG/HDL-C), in-hospital mortality, 28-day survival rate, and 28-day survival time.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* ICU stay ≥24 hours
* ulfillment of the diagnostic criteria for sepsis according to the Sepsis-3 definition, which included:
* (a) suspected or confirmed infection based on clinical evidence and/or positive microbiological findings;
* (b) Sequential Organ Failure Assessment (SOFA) score ≥2 points

Exclusion Criteria:

* cognitive impairment related to sedation
* pregnancy
* inability to communicate effectively due to visual, auditory, or language disorders
* primary central nervous system diseases (e.g., cerebrovascular disease, central nervous system infection, autoimmune encephalitis, or epileptic seizures)
* intolerance or allergy to benzodiazepines, or a history of myasthenia gravis, schizophrenia, or severe depressive disorder
* metabolic encephalopathy (including hypoglycemia, diabetic ketoacidosis, hepatic encephalopathy, pulmonary encephalopathy, or uremic encephalopathy)
* poisoning
* skull fracture or intracranial injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with sepsis in the ICU
Sampling Method: Non-Probability Sample
Enrollment: 2734 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
The incidence of sepsis-associated encephalopathy (SAE) | 3 days
  Glasgow Coma Scale (GCS) score of less than 15 or the presence of delirium symptoms confirmed by the Confusion Assessment Method for the ICU (CAM-ICU)

SECONDARY OUTCOMES:
In-hospital mortality | From hospital admission until discharge or in-hospital death, whichever occurred first, assessed up to 90 days.
  In-hospital mortality will be assessed by reviewing medical records from the time of admission to discharge. Deaths occurring during the hospitalization period will be recorded.
Survival time | 28 days
  Patients will be followed up for 28 days after enrollment, and the survival time and rate within 28 days will be recorded
FBG/HDL-C ratio (fasting blood glucose to high-density lipoprotein cholesterol ratio) | 3rd day
  The FBG/HDL-C ratio will be calculated as a single continuous variable (fasting blood glucose divided by HDL-C). This is a single outcome measure. Record the patient's FBG/HDL-C on the 3rd day.

CONTACTS AND LOCATIONS:
Overall Officials: Shusheng Li, PhD, Principal Investigator — Tongji Hospital
Locations (1):
- Department of Critical Care Medicine, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No